CLINICAL TRIAL: NCT01660334
Title: Special Investigation of Vfend on Scedosporisis
Brief Title: Voriconazole (Vfend) Special Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501077
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-10

CONDITIONS: Scedosporium Infection
Keywords: Systemic Mycosis; Scedosporium infection; Scedosporisis; Japanese; voriconazole; VFEND; Regulatory Post Marketing Commitment Plan.
MeSH Terms: conditions — scedosporiosis | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Voriconazole: Subjects who are treated with voriconazole
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Voriconazole Intravenous Solution 200 mg:
  Voriconazole is administered by intravenous drip infusion at the dose of 6 mg/kg twice daily on day 1 and 3 mg/kg or 4 mg/kg twice daily from day 2 onward in adults.
  Voriconazole Tablet 50 mg/ Voriconazole Tablet 200 mg:
  administration for an adult (weighing 40 kg or more) is voriconazole 300mg orally twice daily between meals for day 1 and then 150 mg or 200 mg twice daily between meals from day 2 onward.
  Depending on the symptoms or in cases where the effect is insufficient, the dosage may be increased.
  However, the maximum dose on day 1 must be 400 mg twice daily, and the maximum dose from day 2 onward must be 300 mg twice daily.
  In patients weighing less than 40 kg, voriconazole 150 mg shall be administered twice daily on day 1, and voriconazole 100 mg shall be administered twice daily from day 2 onward.
  Depending on the symptoms, the maintenance dose from day 2 onward may be increased to 150 mg twice daily.
  Other Names: VFEND for Intravenous Use, Voriconazole for Intravenous Use, VFEND Tablets, Voriconazole Tablet

SUMMARY:
To collect the efficacy and safety information of voriconazole related to their appropriate use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

Male or Female patients who are prescribed voriconazole (VFEND) for deep mycosis on Scedosporisis.

Exclusion Criteria:

Subject who have been prescribed voriconazole (VFEND) for deep mycosis on Aspergillus, Candidasis,Cryptococcal infections not involving Scedosporisis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A1501077 prescribes the voriconazole (VFEND).
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501077&StudyName=Voriconazole%20%28Vfend%29%20Special%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29%20%20%0A%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole for Scedosporium Disease: Participants taking Voriconazole for Scedosporium disease according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Voriconazole for Scedosporium Disease
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole for Scedosporium Disease
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  <65 years | 4
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Voriconazole, irrespective of causal relationship to Voriconazole (including clinically problematic abnormal changes in laboratory test values). Serious adverse events were defined as those including death, fatal risk, hospitalization or prolongation of hospitalization period, continuous dysfunction, those causing malformation, and serious ones like the above-cited events. Treatment related Adverse Events were evaluated in company with the causal relationship to Voriconazole.
Time Frame: 16 weeks
Population: The safety analysis population consists of the participants who satisfy the case conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Voriconazole for Scedosporium Disease
Number analyzed (Participants) | 12
participants | 2

2. Secondary Outcome: Number of Participants With Clinical Response of Cure at the Test-of-Cure(TOC) Visit.
Description: The primary endpoint was the efficacy ratio (number of effective cases/number of evaluable cases for efficacy assessment) among the cohort comprising the participants for efficacy analysis.
  Clinical response of cure was assessed comprehensively by physicians in the three categories, which were "effective", "ineffective", and "not evaluable", based on the clinical symptoms, imaging diagnosis and endoscopy, fungal tests, and serological tests.
Time Frame: 16 weeks
Population: The efficacy analysis population basically consists of the evaluable cases in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Voriconazole for Scedosporium Disease
Number analyzed (Participants) | 11
participants | 6

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study.
Arm/Group | Voriconazole for Scedosporium Disease
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voriconazole for Scedosporium Disease (N=12)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voriconazole for Scedosporium Disease (N=12)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.